CLINICAL TRIAL: NCT05403242
Title: A Multicenter, Open Label，Single Arm，Phase Ib/II Study to Evaluate the Effect and Safety of RC48-ADC Combined With S-1 for First-line Treatment of Advanced Gastroesophageal Adenocarcinoma With Moderate Expression of HER2
Brief Title: RC48-ADC Combined With S-1 for First-line Treatment of Advanced Gastroesophageal Adenocarcinoma With Moderate Expression of HER2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor and chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2022-132-01
Record Dates: First submitted 2022-05-06; First posted 2022-06-03 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Advanced Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC Combined With S-1 (Experimental)
  Interventions: Drug: RC48-ADC; Drug: S-1

INTERVENTIONS:
Drug: RC48-ADC — 2.0 mg/kg, IV, d1, every 2 weeks; or 2.5 mg/kg, IV, d1, every 2 weeks
Drug: S-1 — 40-60 mg, bid po, d1-10, every 2 weeks

SUMMARY:
This study was a single-arm, open, multi-center Phase Ib/II clinical trial to observe and evaluate the efficacy and safety of RC48-ADC plus S-1 in first-line treatment of advanced gastroesophageal adenocarcinoma with moderate expression of HER2.

ELIGIBILITY:
Inclusion Criteria:

* At the same time, patients voluntarily participated in the study and signed informed consent;
* Either male or female, aged 18 or older;
* Patients diagnosed by pathological or cytological diagnosis of gastric cancer (GC), gastroesophageal junction carcinoma (GEJ) or esophageal adenocarcinoma had evidence of local advanced lesions or metastases that could not be surgically resected, and were mostly adenocarcinoma confirmed by histological examination;
* No previous systemic therapy; Or had received neoadjuvant/adjuvant chemotherapy but experienced disease progression or recurrence 6 months after the end of treatment;
* HER2 IHC 2+ and FISH-;
* ECOG scores 0-1;
* Estimated survival ≥3 months;
* Women of reproductive age had to undergo a pregnancy test (serum or urine) which was negative within 7 days of enrollment, and volunteer to use an appropriate method of contraception during the observation period and for 12 weeks after the last study drug was given. For men, surgical sterilization or consent to use appropriate methods of contraception during the observation period and for 12 weeks after the last administration of the study drug;
* Patients who comply are expected to be able to follow up on therapeutic outcomes and adverse reactions as required by the regimen.

Exclusion Criteria:

* Five years before first use of the study drug has been diagnosed as other malignant tumor, the effective treatment of basal cell carcinoma, squamous cell carcinoma of the skin and/or the effective removal of cervical cancer in situ and/or except breast cancer;
* Known hypersensitivity to RC48-ADC;
* HBV DNA>500 IU/ mL (or 2000 copies /ml), HCV RNA>103 copies /ml, HBsAg+ and anti-HCV antibody positive;
* History of HIV infection;
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment;
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxity | through study completion, an average of 1 year
ORR（Objective Response Rate） | Imaging tests were performed every 6 weeks (±7 days) from the first year of treatment to assess efficacy, and every 8 weeks (±7 days) after 1 year
  The proportion of patients whose tumors shrink by a certain amount and remain so for a certain amount of time, including CR+PR cases.

SECONDARY OUTCOMES:
PFS(progression-free survival) | Imaging tests were performed every 8 weeks (±7 days) from the first year of treatment to assess efficacy, and every 7 weeks (±7 days) after 1 year
  Time from randomness to the first occurrence of disease progression or death from any cause.
DOR(Duration of Response ) | Imaging tests were performed every 6 weeks (±7 days) from the first year of treatment to assess efficacy, and every 8 weeks (±7 days) after 1 year
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
OS(Overall Survival) | From date of randomization until the date of death from any cause, assessed up to 24 months
  Time from randomization to death from any cause
AE(Adverse Event) | Up to 2 years
  The drug safety was assessed by investigator(s) according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No